CLINICAL TRIAL: NCT00983697
Title: A Multicenter Trial of FDG-PET/CT Staging of Head and Neck Cancer and Its Impact on the N0 Neck Surgical Treatment in Head and Neck Cancer Patients
Brief Title: FDG-PET/CT in Assessing the Tumor and Planning Neck Surgery in Patients With Newly Diagnosed H&N Cancer
Acronym: ACRIN6685
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000654703; ACRIN-6685 (Other: CIP ID); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG PET/CT (Experimental): Planning for Therapeutic conventional surgery of the N0 neck is documented prior to and immediately after review of the fludeoxyglucose F 18 (FDG)-PET/CT scan completed per protocol.
  Interventions: Procedure: therapeutic conventional surgery; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Procedure: therapeutic conventional surgery
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic procedures, such as fludeoxyglucose F 18-PET/CT scan, may help doctors find head and neck cancer and find out how far the disease has spread. It may also help doctors plan the best treatment.

PURPOSE: This phase II trial is studying fludeoxyglucose F 18-PET/CT imaging to see how well it works in assessing the tumor and planning neck surgery in patients with newly diagnosed head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the negative predictive value of PET/CT imaging based upon pathologic sampling of the neck lymph nodes in patients with head and neck cancer planning to undergo N0 neck surgery.
* Determine the potential of PET/CT imaging to change treatment.

Secondary

* Estimate the sensitivity and diagnostic yield of PET/CT imaging for detecting occult metastasis in the clinical N0 neck (both by neck and lymph node regions) or other local sites.
* Determine the effect of other factors (e.g., tumor size, location, secondary primary tumors, or intensity of FDG uptake) that can lead to identification of subsets of patients that could potentially forego neck dissection or that can provide preliminary data for subsequent studies.
* Compare the cost-effectiveness of using PET/CT imaging for staging head and neck cancer vs current good clinical practices.
* Evaluate the incidence of occult distant body metastasis discovered by whole-body PET/CT imaging.
* Correlate PET/CT imaging findings with CT/MRI findings and biomarker results.
* Evaluate the quality of life of these patients, particularly of those patients whose management could have been altered by imaging results.
* Evaluate PET/CT imaging and biomarker data for complementary contributions to metastatic disease prediction.
* Compare baseline PET/CT imaging and biomarker data with 2-year follow up as an adjunct assessment of their prediction of recurrence, disease-free survival, and overall survival.
* Determine the proportion of neck dissections that are extended (i.e., additional levels that clinicians intend to dissect beyond the initial surgery plan) based on local-reader PET/CT imaging findings shared with the surgeon before dissection.
* Estimate the optimum cutoff value of standardized uptake values for diagnostic accuracy of PET/CT imaging.
* Evaluate the impact of PET/CT imaging on the N0 neck across different tumor subsites (defined by anatomic location).

OUTLINE: This is a multicenter study.

Patients undergo fludeoxyglucose F 18-PET/CT imaging. Approximately 14 days later, patients undergo unilateral or bilateral neck dissection.

Patients complete quality-of-life questionnaires at baseline and at 1, 12, and 24 months after surgery.

Patients undergo blood and tissue sample collection periodically for biomarker analysis.

Patients are followed up periodically for up to 2 years after surgery.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed squamous cell carcinoma (SCC) of the head and neck , including any of the following sites:

  * Oral cavity
  * Oropharynx, including base of tongue and tonsils
  * Larynx
  * Supraglottis
* Stage T2-T4, N0-N3 disease

  * Unilateral or bilateral neck dissection planned

    * No N2c disease (if bilateral disease is present)
  * Has ≥ 1 clinically N0 neck side as defined by clinical exam (physical exam with CT scan and/or MRI)

    * A N0 neck must be planned to be dissected for the patient to be eligible
    * . The N0 neck can be either ipsilateral to the head and neck tumor or the contralateral N0 neck if a bilateral neck dissection is planned
* CT scan and/or MRI taken within the past 4 weeks to confirm SCC of the head and neck

  * Simultaneous diagnostic CT with PET scan allowed; however, PET cannot be used as part of the criteria to define the N0 neck disease
  * For CT scan and/or MR images from other institutions, ACRIN recommends a re-read by a local neuro-radiologist to ensure compliance
* No sinonasal cancer, salivary gland cancer, thyroid cancer, nasopharyngeal cancer, or advanced skin cancer

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Weight ≤ 350 lbs
* No poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL) despite attempts to improve glucose control by fasting duration and adjustment of medications (optimally, patients will have glucose < 150 mg/dL)
* No underlying medical condition that would preclude surgery (neck dissection)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2010-04-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of PET/CT imaging for staging the N0 neck based upon pathologic sampling of the neck lymph nodes | Within Two Weeks Before Surgery and after sampling of neck lymph nodes
  True negative cases will be determined by histopathology reports. The test will be defined as positive when SUVmax value of ≥ 2.0; and negative otherwise.

SECONDARY OUTCOMES:
Sensitivity and diagnostic yield of PET/CT imaging for detecting occult metastasis in the clinically N0 neck (both by neck and lymph node regions) or other local sites | Within Two Weeks Before Surgery and after sampling of neck lymph nodes
  True positive cases will be determined by histopathology reports. The test will be defined as positive when SUVmax value of ≥ 2.0; and negative otherwise. The diagnostic yield is defined as the ratio of cancers to total screened
Determine which factors (e.g., tumor size, secondary primary tumors, location, or intensity of FDG uptake) may identify patients who can forego neck dissection | Within Two Weeks Before Surgery and after sampling of neck lymph nodes
  True positive cases will be determined by histopathology reports. The test will be defined as positive when SUVmax value of ≥ 2.0; and negative otherwise. The diagnostic yield is defined as the ratio of cancers to total screened
Cost-effectiveness and cost-benefit of using PET/CT imaging for staging of head and neck cancer vs current good clinical practices | 2 years post-surgery
  The outcome measure will use the total cost of care for each participant to compute the incremental cost-effectiveness ratio (ICER)
Incidence of occult distant body metastasis discovered by whole body PET/CT imaging | Within Two Weeks Before Surgery
  this outcome will count the distant body metastasis not previously seen and report the results as a percentage.
Correlation of PET/CT imaging findings with CT/MRI findings and biomarker results | Within Two Weeks Before Surgery
  the outcome measure will consist of paired proportions of dichotomized PET/CT and CT/MRI test results; and biomarker test results
Quality of life (QOL), particularly in patients whose management could have been altered by imaging results | 2 years post-surgery
  QOL will be assessed using SF-36, Non-Utility HUI, and UW-QoL scores
Evaluation of the PET/CT imaging and biomarker data for complementary contributions to metastatic disease prediction | Within Two Weeks Before Surgery
  the metastatic disease status is the response variable and PET/CT test results and biomarker data are predictors.
Comparison of baseline PET/CT imaging and biomarker data with 2-year follow up as an adjunct assessment of their prediction of recurrence | 2 years post-surgery
  model the associations of PET/CT test results and biomarker data (predictors) to recurrence
Comparison of baseline PET/CT imaging and biomarker data with 2-year follow up as an adjunct assessment of their prediction of disease-free survival | 2 years post-surgery
  model the associations of PET/CT test results and biomarker data (predictors) to disease-free survival
Comparison of baseline PET/CT imaging and biomarker data with 2-year follow up as an adjunct assessment of their prediction of overall survival | 2 years post-surgery
  model the associations of PET/CT test results and biomarker data (predictors) to overall survival (censored responses)
Proportion of neck dissections that are extended based on local-reader PET/CT imaging findings shared with the surgeon before dissection | Within Two Weeks Before Surgery
  Outcome is defined as the number patients who surgeons intend to dissect levels beyond the initial surgery plan
Optimum cutoff value of standardized uptake values for diagnostic accuracy of PET/CT imaging | Within Two Weeks Before Surgery
  ROC analysis will be used to maximize the youden index and estimate the optimum cutoff value of SUV for diagnostic accuracy of PET/CT on N0 neck
Impact of PET/CT imaging on the N0 neck across different tumor subsites (defined by anatomic location) | Within Two Weeks Before Surgery
  Diagnostic Accuracy measures will be calculated using ROC analysis, subset by anatomic location

CONTACTS AND LOCATIONS:
Overall Officials: Val J. Lowe, MD, Study Chair — Mayo Clinic
Locations (12):
- United States (11):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Morton Plant Mease Cancer Care at Mease Countryside Hospital, Safety Harbor, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Jewish Hospital Heart and Lung Institute, Louisville, Kentucky
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
See ACRIN data sharing policy:
  https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx
Time Frame: by request 6+ mo after publication available through The Cancer Imaging Archive expected 1-year after publication.
Access Criteria: Safe-Harbor deidentified data

REFERENCES:
- [Result] Lowe VJ, Duan F, Subramaniam RM, Sicks JD, Romanoff J, Bartel T, Yu JQM, Nussenbaum B, Richmon J, Arnold CD, Cognetti D, Stack BC Jr. Multicenter Trial of [18F]fluorodeoxyglucose Positron Emission Tomography/Computed Tomography Staging of Head and Neck Cancer and Negative Predictive Value and Surgical Impact in the N0 Neck: Results From ACRIN 6685. J Clin Oncol. 2019 Jul 10;37(20):1704-1712. doi: 10.1200/JCO.18.01182. Epub 2019 Feb 15. PMID 30768363
- See also: National Cancer Institute's clinical trials database — https://clinicaltrials.gov/ct2/show/NCT00983697